CLINICAL TRIAL: NCT00589745
Title: Measurement of Transepithelial Nasal Potential Difference (NPD) for the Diagnosis of Cystic Fibrosis
Brief Title: Nasal Potential Difference (NPD) for the Diagnosis of Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-001589
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis
Keywords: Diagnosis
MeSH Terms: conditions — Cystic Fibrosis; Disease | interventions — neodymium pyrocatechin disulfonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects being evaluated for CF (Other): Subjects will be referred from physicians who are clinically concerned about the possibility of Cystic Fibrosis. Nasal potential difference measurement will be obtained to potentially help aid in diagnosis.
  Interventions: Other: Nasal potential difference measurement

INTERVENTIONS:
Other: Nasal potential difference measurement — Nasal potential difference measurement involves dripping small amounts of 5 test solutions into the anterior nostril. This is designed to test the ability of the cells to regulate the movement of salt and water in people with features of CF in whom the diagnosis is not entirely clear.
  Other Names: NPD

SUMMARY:
The purpose of this research study is to provide a novel method for the diagnosis of Cystic Fibrosis (CF). This protocol is designed to test the ability of the cells to regulate the movement of salt and water in people with features of CF in whom the diagnosis is not entirely clear. We will be studying these cells in the nose, by a technique called nasal transepithelial potential difference (NPD).

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is an autosomal recessive systemic disorder of exocrine glands and secretory epithelia. The disease results from mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene which cause a variety of abnormalities. CFTR is absent or dysfunctional in cystic fibrosis. Most of the defects in CFTR result in abnormal chloride ion transport and abnormally viscous mucus. Nasal epithelial CFTR function will be assessed by the NPD procedure.

NPD measurements are useful as a diagnostic tool in individuals with borderline or normal sweat chlorides, one or no identified CFTR mutations, and a clinical history suggestive of CF. The NPD has become the gold standard for detection and quantification of CFTR function in the airways. The assay has also served as an important endpoint since 1981. It has been used extensively and is standardized to assess the ability of new therapeutics in studies designed to replace, repair or restore defective ion transport in CF patients.

The assay basically involves dripping small amounts of the test solutions into the anterior nostril in order to measure uptake or secretion of sodium and chloride. There are five solutions required for the NPD measurement:

* Solution #1: Buffered Ringers
* Solution #2: Solution #1+Amiloride
* Solution #3: Buffered Zero Chloride Solution + Amiloride
* Solution #4: Solution #3 + Isoproterenol
* Solution #5: Solution #4 + Adenosine 5'-Triphosphate-Disodium salt (ATP)

The Cystic Fibrosis Therapeutics Development Network (TDN) is a formal affiliation of CF Research Centers in the US. Two Standard Operating Procedures have been developed by the TDN for the NPD procedure and qualification of those performing the measurement.

Procedure Details:

Briefly, a series of stopcocks is configured to allow perfusion of the above solutions through the port at the tip of an exploring catheter (PE50 tubing. All test solutions are perfused at a rate of 5.0 cc per minute. In each nostril, the PD readings in Ringer's at 0.5, 1.0, 1.5, 2, and 3 cm (lumen negative) are averaged and taken as the average 'baseline' PD. The catheter tip is then placed at the most negative PD site and maintained for superperfusion measurements with a small piece of tape applied to the nasal tip (to hold the catheter for the duration of the protocol). All solutions are warmed to 37˚C prior to contact with the nasal mucosa.

For each perfusion condition, a steady-state recording is obtained. The recording lasts at least one minute (for Solution #1) and for three minutes (for Solutions #2, 3, and 4) prior to proceeding to the next solution within the sequence. Solution #5 is perfused for a minimum of one minute, and confirms retention of ATP-activated Clˉ secretion in both CF and non-CF individuals. Several readings are obtained for data analysis, and then all nasal P.D. tracings are scored by investigators.

ELIGIBILITY:
Inclusion Criteria:

* All ethnic groups accepted
* Individuals with borderline or normal sweat chloride, one or no identified CFTR mutations and a clinical history suggestive of CF.
* Children less than 6-8 years of age may be unable to cooperate (hold still) for the procedure, or be frightened by the procedure. Sedation may be necessary for performance of the procedure on a young child

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-09; Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
The basis of analysis will be the NPD response patterns, which will be interpreted and classified by the PI, as consistent or inconsistent with the diagnosis of CF based on comparison with published standards. | Every visit

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Rubenstein, M.D., PhD., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States